CLINICAL TRIAL: NCT04914585
Title: Automatic Optical Identification of the Spine Vertebrate Using Three-dimensional Optical Detection Based on a CT Test
Status: Recruiting | Type: Observational
Sponsor: Deep Health Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 0001 (IRB 0485-19)
Record Dates: First submitted 2021-05-30; First posted 2021-06-04 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-06

CONDITIONS: Spinal Surgery of Vertebrae, Intervertebral Discs and the Spinal Cord; CT Scans
Keywords: spinal surgery; CT scans; surgical navigation; optical tracking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
CT scans of the spine include vertebrae, intervertebral discs and the spinal cord. These tests are performed in an orderly protocol and allow for three-dimensional reconstruction of the vertebra in sagittal and coronal guides.

DETAILED DESCRIPTION:
In spinal surgery, there are a number of navigation technologies based on CT scans performed before surgery (or during surgery) and identify the vertebrae (using special photographs or markers on the spine), such as Mazor with the Renaissance Robotic Surgical System used in hospitals, or BrianLab Which uses non-robotic navigation and is based on a marker located on the patient's back. These technologies are not optimal, and have a number of significant drawbacks: Because during spinal surgery, there is a displacement, the level of accuracy decreases as the surgery progresses. In addition, there is extensive use of radiation in these means since in many cases CT is performed before and during surgery.

Today, in the age of optical detection, it is possible to detect three-dimensional structures in photography and allow high levels of accuracy (less than 0.5 mm). Optical scanning does not include radiation and lasts the entire length of the operation. Of the patient and of the treating staff.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* 18 and above years old
* Patients who have available spinal CT tests will be included in the study
* Patients who are about to undergo spinal surgery

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidates for spinal surgery in the Orthopedics department at Hadassah medical center who have a previous CT scan of the spine. The participant will receive an explanation and will undergo a process of informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
DEEP HEALTH's detection algorithm for optical detection of vertebrae in the spine in patients undergoing spinal surgery. | 12 months
  Verify an algorithm for automatic detection of vertebrae in the spine, while building an optical model for optical identification in the operating room, and reducing the need for radiation use during spinal surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Josh Schroeder, MD, Principal Investigator — Advisor
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farah K, Coudert P, Graillon T, Blondel B, Dufour H, Gille O, Fuentes S. Prospective Comparative Study in Spine Surgery Between O-Arm and Airo Systems: Efficacy and Radiation Exposure. World Neurosurg. 2018 Oct;118:e175-e184. doi: 10.1016/j.wneu.2018.06.148. Epub 2018 Jul 3. PMID 30257292
- [Background] Gebhard F, Weidner A, Liener UC, Stockle U, Arand M. Navigation at the spine. Injury. 2004 Jun;35 Suppl 1:S-A35-45. doi: 10.1016/j.injury.2004.05.009. PMID 15183702
- [Background] Mendelsohn D, Strelzow J, Dea N, Ford NL, Batke J, Pennington A, Yang K, Ailon T, Boyd M, Dvorak M, Kwon B, Paquette S, Fisher C, Street J. Patient and surgeon radiation exposure during spinal instrumentation using intraoperative computed tomography-based navigation. Spine J. 2016 Mar;16(3):343-54. doi: 10.1016/j.spinee.2015.11.020. Epub 2015 Dec 10. PMID 26686604